CLINICAL TRIAL: NCT02608164
Title: A Comparison of Capsules and Oral Spray Solution as Methods of Delivering Vitamin D3 and Raising Status: a Randomised Crossover Study
Brief Title: A Comparison of Capsules and Oral Spray Solution as Methods of Delivering Vitamin D3 and Raising Status
Acronym: SCD3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Northern Ireland Executive (Unknown); HSC Public Health Agency (Unknown)
Responsible Party: Principal Investigator, Dr Pamela Magee, Dr Pamela Magee, University of Ulster
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: REC/15/0083
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Vitamin D Concentration; Vitamin D Status
Keywords: Healthy adults
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D oral spray solution (Active Comparator): An oral spray solution containing 3000IU (75micrograms) vitamin D3 per spray
  Interventions: Dietary Supplement: 3000IU(75μg) vitamin D3
- Vitamin D capsules (Active Comparator): A capsule containing 3000IU (75micrograms) vitamin D3 per capsule
  Interventions: Dietary Supplement: 3000IU(75μg) vitamin D3

INTERVENTIONS:
Dietary Supplement: 3000IU(75μg) vitamin D3
  Other Names: cholecalciferol

SUMMARY:
The aim of the study is to compare the effectiveness of a vitamin D3 oral spray solution with capsules at raising vitamin D status over winter.

This randomised crossover trial will aim to recruit a total of 22 healthy participants for a total of two 4-week interventions separated by a 10-week washout.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy
* Over the age of 18

Exclusion Criteria:

* Those that intend to consume a supplement containing vitamin D at any point during the study
* Those under the age of 18.
* Individuals that are on prescribed medication that is known to affect vitamin D metabolism
* Those following a vegan diet
* Sun-bed users
* Participants that are planning a sun holiday during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Total 25-hydroxyvitamin D concentration | At baseline and weeks 4, 14 and 18
  Total 25-hydroxyvitamin D concentration will be determined using liquid chromatography-tandem mass spectrometry in collected serum samples

SECONDARY OUTCOMES:
Biomarkers of vitamin D metabolism | At baseline and weeks 4, 14 and 18
  Biomarkers of vitamin D metabolism, including parathyroid hormone and adjusted calcium will be quantified in collected serum samples by ELISA and using a clinical chemistry analyser
Dietary vitamin D intake | At week 18 only
  Dietary vitamin D and calcium intake will be estimated using a validated food frequency questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pamela J Magee, PhD, Principal Investigator — University of Ulster
Locations (1):
- Human Intervention Studies Unit (HISU), University of Ulster, Coleraine, Londonderry, United Kingdom